CLINICAL TRIAL: NCT06739642
Title: Effectiveness of Caregiver Nutrition Education on the Diet of Patient with Dementia: a Randomized Controlled Trial
Brief Title: Effectiveness of Dementia Nutrition Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Fatma Uyar Açışlı, Phd, Manisa Celal Bayar University, Public Health Nursing Department, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CBU-NURS-FUA-01
Record Dates: First submitted 2024-12-05; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Dementia; Nutrition; Nutrition Deficiency Due to Insufficient Food; Nutrition Assessment
Keywords: Dementia, Caregiving, Nutrition and Feeding Issues, Education and Training, Nursing.
MeSH Terms: conditions — Dementia | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): caregivers in the intervention group (n=45) received an individualized educational program intervention
  Interventions: Other: Education
- Control (No Intervention): Caregivers in the control group (n=44) continued to receive routine care.

INTERVENTIONS:
Other: Education — caregivers in the intervention group received an individualized educational program intervention. The content of the educational program was developed by the researcher through a review of the literature and interviews with caregivers. The educational program, during three months, was delivered in 6 sessions of 40 minutes each. The topics of the training content were as follows: 1. General Nutrition Information, 2. Changes Affecting Nutrition During Old Age and Nutrition Principles, 3. Anthropometric Measurements and Scans, 4. Nutritional Problems in the Patient with Dementia, Dementiamendations for Increasing Nutritional Intake in Dementia Patients, 6. Alternatives for Severe Feeding Problems. Covering general topics was held as group education; carried out in two separate groups. Another individual session was planned for caregivers who could not attend the group education program, and the missing topics were completed.
  Arms: Intervention

SUMMARY:
Nutritional problems can and do manifest themselves at various stages and with varying degrees of severity. Patients with dementia are at significant risk for weight loss and malnutrition due to the numerous issues that arise during the disease process. Caregivers of patients with dementia face significant challenges in providing nutritional care for their patients due to difficulties with nutrition for physical, emotional, cognitive, and behavioral reasons.

The following methods were used: This study employed a randomized controlled trial with a pretest-posttest design. The study was conducted with 89 patients and caregivers (45 in the intervention group and 44 in the control group). We collected data from the intervention and control groups before and after the intervention using the Descriptive Information Form, Edinburgh Nutrition Evaluation in Dementia (EdFED) Scale, Mini Nutritional Assessment, Dysphagia Assessment Scale in Multiple Sclerosis, and Sarcopenia Screening Test (SARC-F). The intervention group received a standardized educational program for three months. We evaluated the data using percentages, arithmetic means, standard deviations, medians, and interquartile ranges. We analyzed the data using chi-square tests, Mann-Whitney U tests, Wilcoxon signed-rank tests, and intention-to-treat analyses.

ELIGIBILITY:
Inclusion criteria for caregivers

* being a primary caregiver,
* aged> 18,
* volunteering to participate in the study.

Exclusion criteria for caregivers -wanting to quit working, not attending training

Inclusion criteria for patients

* According to DSM-V criteria, they must have a nutritional disorder, metabolic disorder, or dementia that is not due to systematic diseases
* be fed orally
* have the caregiver/guardian of the patient with dementia voluntarily agree to participate in the research with him/herself and the patient

Exclusion criteria for patients

-Having a health condition that affects nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
The Edinburgh Nutrition Assessment in Dementia ( EdFED ) Scale | Four months
  The Edinburgh Nutrition Assessment in Dementia ( EdFED ) Scale developed by Watson (Watson, 1994)helps screen for feeding difficulties in patients with dementia. The scale establishes the behavioural baseline and defines the level of assistance the patient needs. Administration of the scale takes less than five minutes. The first 10 items in the scale address feeding behaviour at meals; Depending on how often each behavior occurs during a feeding, 0 points are given for "never", 1 point is given if it occurs 2 or 3 times a week / "sometimes", and 2 points are given if it occurs more than 4 times a week / " often". The score from the first 10 items ranges from 0 to 20, with 20 being the most serious condition. Points can be used to track change. Finally, item 11 states the level of support the patient needs. The scale was reported to be valid and reliable (Cronbach Alpha coefficient = 0.86) (Uyar et al., 2022). In this study, the Cronbach Alpha coefficient was found to be 0.90 in
Dysphagia Assessment Scale in Multiple Sclerosis (DYMUS) | Four months
  Dysphagia Assessment Scale in Multiple Sclerosis (DYMUS) was developed by Bergamaschi et al. (2008) for the evaluation of oropharyngeal dysphagia in patients with Multiple Sclerosis (Bergamaschi et al., 2008). In the scale, the dysphagia score for solids is calculated by adding the 1st, 3rd, 4th, 5th, 7th, 8th and 10th items, and the dysphagia score for liquids is calculated by adding the 2nd, 6th and 9th items. Scale items are coded as "No = 0" and "Yes = 1". Scores between 0 and 10 can be obtained from the scale. A score of 1 or above indicates the presence of dysphagia, and a score of 3 or more indicates the presence of severe dysphagia. Turkish validity and reliability study was conducted by Tenekeci et al. and it has been reported that the total scale of Cronbach's Alpha coefficient has been 0.91 (Tenekeci et al., 2018). In this study, the Cronbach Alpha coefficient was in the pre-test 0.85; it was in the post-test 0.86. Although the scale was developed for patients with MS, app
The Mini Nutritional Assessment (MND) Test | Four months
  The Mini Nutritional Assessment (MND) Test was developed in 1994 in collaboration between the University of TOULOUSE, New Mexico Medical School and Nestle Research Center (Switzerland). MND is widely used in community clinical practice to examine the nutritional status of the elderly and dementia patients. The test consists of 18 items covering anthropometric measurements, dietary behaviours, and global and subjective factors. Malnutrition Indicator Score (MGP) is calculated by summing the preliminary evaluation score and the comprehensive evaluation score. Malnutrition Indicator Score (MGP) can be at least 0 and at most 30. The range of 24-30 points indicates no risk of malnutrition, the range of 17-23.5 points indicates the risk of malnutrition, and scores less than 17 indicate the presence of malnutrition. Mini Nutritional Assessment (MND) is a common screening tool (Guigoz, 2006). Cronbach's alpha coefficient was reported as 0.65 in elderly people with early-stage dementia (Holm &
The Sarcopenia Screening Test (SARC-F) | Four months
  The Sarcopenia Screening Test (SARC-F) was developed as a possible rapid diagnostic test for (Malmstrom & Morley, 2013) questions the individual's assistance needed for weight bearing, walking, getting up from a chair/bed, climbing stairs, and the experience of falling. Scores range from 0 to 10, with 0-2 points for each component. The 0-3 points range represents healthy, and 4 points and above represent sarcopenia and poor outcomes. Its suitability for the geriatric population in Turkey was checked by Kış and Karaca (2021) (Cronbach Alpha coefficient = 0.60) (Kış & Karaca, 2021). In this study, the Cronbach Alpha coefficient was in the pre-test 0.79; it was in the post-test 0.76.
BMI | Four months
  In this study, BMI was used to evaluate the nutritional status of the patient with dementia. In a similar study (Salva et al., 2011) in the literature on the nutrition of dementia patients, weight was monitored by mail. Care was taken to ensure that the measurements were made by the instructions and by the same person.

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, YUNUSEMRE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data may be shared with individual researchers upon request after the study has been completed and published; however, for data security reasons, sharing the data before publication is not being considered.